CLINICAL TRIAL: NCT05213702
Title: A Randomized Controlled Trial to Evaluate the Efficacy and Safety of Automated Needle Targeting (ANT-X) System Compared to Traditional Free Hand Puncture for Renal Access in Percutaneous Nephrolithotomy (PCNL) Performed by Urologists in Training.
Brief Title: A RCT to Evaluate the Efficacy and Safety of Automated Needle Targeting (ANT-X) System Compared to Traditional Free Hand Puncture for Renal Access in Percutaneous Nephrolithotomy (PCNL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Collaborators: NDR Medical Technology Pte Ltd (Industry)
Responsible Party: Principal Investigator, Dr. Yeoh Wei Sien, Doctor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NDR-CT0023
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Male/non-pregnant female subjects between age 18-75 years, both inclusive, who will undergo Percutaneous Nephrolithotomy (PCNL).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional free hand puncture for renal calyx access (Active Comparator): For human PCNL, we target 60 cases of PCNL, 30 ANT-X puncture and 30 traditional free hand puncture performed by 4 urologic trainees(15 cases per urologic trainee).
  Interventions: Device: Renal Calyx punture with traditional free hand or ANT-X device
- RObotic ANT-X device puncture for renal calyx access (Active Comparator): For human PCNL, we target 60 cases of PCNL, 30 ANT-X puncture and 30 traditional free hand puncture performed by 4 urologic trainees(15 cases per urologic trainee).
  Interventions: Device: Renal Calyx punture with traditional free hand or ANT-X device

INTERVENTIONS:
Device: Renal Calyx punture with traditional free hand or ANT-X device — ANT-X device is a software-controlled automated electromechanical arm. It is developed to provide needle guidance for surgeon in MIS. This aims to reduce the surgery time taken and also minimize the radiation withstand by both surgeon and patient. ANT-X device is actually a Delta parallel robot implementing inverse kinematics to achieve effector's movement. Parallel structures excel in their great stiffness and high positioning accuracy. Most of the main components of ANT-X robot are made up of medical grade Polyether ether ketone (PEEK) material. PEEK is preferred to build the robot because it is radiolucent and lightweight while being able to provide relatively high material strength. The device is intended for use together with C-arm fluoroscope (fluoroscopy/CT technology). The fluoroscopy technology is used to provide image guidance for the needle

SUMMARY:
Objectives: This study aims to determine if the device provides an advantage over traditional free hand puncture by comparing the number of attempts required to obtain access, time to achieve access, radiation exposure to patient and surgeon; and complications.

DETAILED DESCRIPTION:
This is a single centre, participant randomized, open label study to evaluate the efficacy and safety of automated needle targeting (ANT-X) system compared to traditional free hand puncture for achieving renal access in Percutaneous lithotomy (PCNL) performed by urologists in training.

Prior to performing kidney puncture on patients, all participating surgeons will undergo a simulation using Medical Simulation 12 balls phantom device with and without use of the ANT-X. Four urologic trainees (with similar little previous PCNL experience) will be recruited for the simulation. Two end points will be assessed: Number of attempts to achieve desired renal puncture and total fluoroscopy time.

This simulation via 12 balls phantom device will involve fluoroscopic screening of calyx and successful puncture by urologic trainees under consultant supervision. Trainees will have 30 attempts of free hand puncture and 30 attempts using the ANT-X. The trainee will only move on to patient's renal puncture once they are able to achieve more than 80% of satisfactory renal puncture on simulator.

For human renal puncture, we will aim for 60 cases of PCNL, 30 to be done using ANT-X puncture and 30 using traditional free hand puncture performed by 4 urologic trainees (15 cases per urologic trainee).

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to sign informed consent form before initiation of any study specific procedures.
* Subjects diagnosed with kidney stones and planned for prone PCNL.
* Male/ non- pregnant female subjects between 18-75 years (both inclusive) of age at the time of informed consent.
* Subjects with renal stones of ≥1 cm or not managed by other stone treatments (e.g. shock wave lithotripsy, ureteroscopy).
* Serum creatinine of < 1.2 mg/dl.

Exclusion Criteria:

* Subjects with bleeding disorders.
* Recent infection of the kidney or urinary tract which leads to pus accumulation in the kidney, i.e., Pyonephrosis.
* Subjects not able to have prone positions for surgical procedure due to comorbid conditions.
* Renal stones < 1 cm and can managed by another technique.
* Patients with moderate to severe renal failure.
* Patients with congenital urinary tract anomalies.
* Patients on anticoagulation or antiplatelet therapy.
* Evidence or history of any other disease that in the opinion of the investigator would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbated during the study.
* Legal incapacity or other circumstances that render the subject unable to understand the nature, scope and possible consequences of the study.
* Clinically significant abnormal findings or condition (other than kidney stone), which might, in the opinion of the Investigator, interfere with study evaluations or pose a risk to subject safety during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-25 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of attempts required to obtain access | Day 0 surgery
  An access attempt is defined as each separate passage of the needle into the kidney. Number of attempts by Investigator/surgeon will be recorded.
Time for the access | Day 0 surgery
  Time to successful access into the collecting system will be calculated in minutes starting from the placement of the needle on the skin surface to the identification of urine efflux from the end of the needle or reach of target. Start time of needle placement and time of urine efflux from the end of the needle or reach of target will be recorded in subject CRF in hh:mm:ss format.

SECONDARY OUTCOMES:
Radiation exposure to patient and surgeon | Day 0 surgery
Assessment of AEs | Admission day till discharge within 7 days
  Advere events associated with the procedure

CONTACTS AND LOCATIONS:
Overall Officials: WS Yeoh, MD, Principal Investigator — UMMC

IPD SHARING:
Plan to Share IPD: No